CLINICAL TRIAL: NCT05631821
Title: Three-axis Correction of Spinal Deformity and Post-implantation Rod Contour Changes Utilizing Differential Rod Bending and Pre-operative Templating in Adolescent Idiopathic Scoliosis: A Pilot Study
Brief Title: 3-D Correction of Adolescent Idiopathic Scoliosis (AIS) With Differential Metals
Acronym: AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Stryker Spine (Industry)
Responsible Party: Principal Investigator, Christopher J DeWald, Director of Spinal Deformity, Rush University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIS Pilot Study
Record Dates: First submitted 2015-05-18; First posted 2022-11-30 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Juvenile and Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Intervention Model Description: Twenty (20) patients prospective and Twenty (20) retrospective. Retrospective matched cohort of patients from the investigating surgeon. The patients will have had surgery using rods but without the MESA™ Spinal Fixation System. The prospective patient will have surgery using rods with the MESA™ Spinal Fixation System.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective Range Spinal System (Active Comparator): Adolescent (between the ages of 10-18 years of age), with Idiopathic Scoliosis Range Spinal System: rod contour changes utilizing Differential Rod Bending and pre-operative templating in Adolescent Idiopathic Scoliosis: A pilot study. The prospective arm consented subjects will use the Rod Counour measurement system
  Interventions: Procedure: differential rod bending with rod contours (MESA Spinal System)
- Retrospective (No Intervention): Retrospective matched cohort of subjects from the investigating surgeon are subjects that have not used the Rod contour measurement system. There is no intervention because the second arm is retrospective chart review.

INTERVENTIONS:
Procedure: differential rod bending with rod contours (MESA Spinal System) — differential rod bending with rod contours and Mesa Spinal system evaluate the correction of adolescent idiopathic scoliosis deformity achieved utilizing a technique of differential rod bending with rod contours pre-operatively determined from a best-fit measure utilizing a computer-based software tool
  Other Names: MESA Spinal System
  Arms: Prospective Range Spinal System

SUMMARY:
This study is designed to evaluate the coronal, sagittal, and axial correction of deformity secondary to adolescent idiopathic scoliosis utilizing a technique employing a posterior spinal fusion construct utilizing rods of different material rigidity and asymmetric bends determined using computer-based software to pre-operatively template a best-fit rod contour from pre-operative radiographs. To further evaluate the changes in contour of the rods from the pre-operative templates to the post-implantation radiographs.

DETAILED DESCRIPTION:
Current posterior instrumentation devices employ pedicle screw and hook based systems to correct spinal deformity. Challenges remain for surgeons to appropriately contour the rods used to achieve the desired correction. The current practice is for the surgeon to intra-operatively contour the rod using various bending tools based on the appearance of the spine. The surgeon visually estimates the amount of bend needed and contours the rod accordingly. Changes in rod contours during implantation from the forces of correction limit the ability to achieve desired and optimal corrections. This is possibly related to both inaccurate bending estimates as well as techniques that affect the peri-implantation rod contours. These phenomena may lead to complications including but not limited to failure of hardware, coronal and/or sagittal spinal imbalance, and adjacent segment pathology or failure. The ability for the surgeon to pre-operatively calculate the proper bends to generate a predictable correction may improve patient outcomes by achieving better overall correction, better coronal and sagittal balance, reduce adjacent segment pathology.The purpose of this study is to evaluate the correction of adolescent idiopathic scoliosis deformity achieved utilizing a technique of differential rod bending with rod contours pre-operatively determined from a best-fit measure utilizing a computer-based software tool,Surgimap Spine to generate a template for manual rod contouring. The study will correlate the post-operative changes in rod contours with the correction achieved in spinal deformity. The pilot study will be used to validate the model for a prospective, randomized, multi-center, study of statistical power to compare the results of pre-operatively determined rod contours to intra-operatively determined rod contours

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of adolescent idiopathic scoliosis. Qualified patients will be confirmed for inclusion by patient history and radiographic studies
2. Lenke Classification Curve type 1, 2, or 3.
3. Willing and able to comply with the requirements of the protocol including follow-up requirements
4. Willing and able to sign a study specific informed consent
5. Skeletally mature (Risser grade III or higher, closed tri-radiate cartilage) between the ages of 10 and 18 years of age

Exclusion Criteria:

1. Previous spine surgery
2. Previous posterior spine surgery (e.g., posterior decompression) that destabilizes the lumbar spine
3. Active systemic infection or infection at the operative site
4. Co-morbid medical conditions of the spine or upper/lower extremities that may affect the lumbar spine neurological and/or pain assessment
5. Metabolic bone disease such as osteoporosis and osteopenia that contraindicates spinal surgery
6. History of an osteoporotic fracture
7. History of an endocrine or metabolic disorder (e.g., Paget's disease) known to affect bone and mineral metabolism
8. Taking medications that may interfere with bony/soft tissue healing including chronic steroid use
9. Known allergy to titanium or cobalt chrome
10. Rheumatoid arthritis or other autoimmune disease or a systemic disorder such as HIV, active hepatitis B or C, or fibromyalgia
11. Insulin-dependent type 1 or type 2 diabetes
12. Medical condition (e.g., unstable cardiac disease, cancer) that may result in patient death or have an effect on outcomes prior to study completion
13. Pregnant, or intends to become pregnant, during the course of the study
14. Severe obesity (Body Mass Index > 40)
15. Physical or mental condition (e.g., psychiatric disorder, dementia, Alzheimer's disease, alcohol or drug addiction) that would interfere with patient self-assessment of function, pain, or quality of life.
16. Involved in current or pending spinal litigation where permanent disability benefits are being sought
17. Incarcerated at the time of study enrollment
18. Current participation in an investigational study that may impact study outcomes
19. Lenke Classification Curve Type 4, 5, or 6.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Pre-op and Post-op Standing Coronal Spinal Xrays | 24 months
  Standard Radiographic Cobb Measurements in degrees in Coronal view

SECONDARY OUTCOMES:
Pre-op and Post-op Standing Sagittal Spinal Xrays | 24 months
  Standard Radiographic Cobb Measurements in degrees in Sagittal view

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J DeWald, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cidambi KR, Glaser DA, Bastrom TP, Nunn TN, Ono T, Newton PO. Postoperative changes in spinal rod contour in adolescent idiopathic scoliosis: an in vivo deformation study. Spine (Phila Pa 1976). 2012 Aug 15;37(18):1566-72. doi: 10.1097/BRS.0b013e318252ccbe. PMID 22426445
- [Result] Luk KD, Vidyadhara S, Lu DS, Wong YW, Cheung WY, Cheung KM. Coupling between sagittal and frontal plane deformity correction in idiopathic thoracic scoliosis and its relationship with postoperative sagittal alignment. Spine (Phila Pa 1976). 2010 May 15;35(11):1158-64. doi: 10.1097/BRS.0b013e3181bb49f3. PMID 20118836